CLINICAL TRIAL: NCT01824446
Title: A Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [14C]SSP-004184 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: AME (Absorption, Metabolism, and Excretion) of Radiolabeled SSP-004184
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SPD602-109
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Healthy
MeSH Terms: interventions — 4,5-dihydro-2-(2-hydroxy-3-(3,6,9-trioxadecyloxy)phenyl)-4-methyl-4-thiazolecarboxylic acid

ARMS (1):
- Radiolabeled SPD602 (Experimental)
  Interventions: Drug: Radiolabeled SPD602 (FBS0701, SSP-004184)

INTERVENTIONS:
Drug: Radiolabeled SPD602 (FBS0701, SSP-004184) — A single oral dose of 3g of radio-labelled SSP-004184 on Day 1
  Other Names: SPD602

SUMMARY:
To evaluate how the body absorbs, metabolizes (breaks down) and excretes (eliminates) the study drug. Further, the study will determine how much of the study drug gets into the bloodstream and how long it takes the body to get rid of it when given as a single dose to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male subjects aged between 18 and 65 years inclusive

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2013-05-29 (Actual); Study Completion 2013-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Covance Clinical Research Unit Inc, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- [14C]SSP-004184: A single oral dose of 3g of radio-labelled SSP-004184 on Day 1
Period: Overall Study
Arm/Group | [14C]SSP-004184
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.2 (3.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 6

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC 0→∞) of Radiolabelled SSP-004184
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Within 30 minutes pre-dose, and Post-dose 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, & 288 hours.
Population: The Pharmacokinetic Analysis Set (PAS) was defined as all subjects in the Safety Analysis Set (SAS) for whom the primary pharmacokinetic data are considered sufficient and interpretable. The SAS consisted of subjects who received at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
ng*hr/ml | 251438.3 (59522.8)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Radiolabelled SSP-004184
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
ng/ml | 119000.0 (35014.3)

3. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Radiolabelled SSP-004184
Description: Tmax is the time after administration of a drug when the maximum plasma concentration in the body is reached.
Time Frame: as for outcome 1
Population: PAS
Measure: Median (Full Range); unit: hours
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
hours | 1.0 [1.0 to 1.5]

4. Primary Outcome: Plasma Half-Life (T1/2) of Radiolabelled SSP-004184
Description: The time it takes for the blood plasma concentration of a substance to halve.
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
hours | 13.039 (5.061)

5. Primary Outcome: Total Body Clearance (CL/F) of Radio-Labelled SSP-004184
Description: The rate at which a drug is removed from the body.
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
L/hr | 12.754 (4.251)

6. Primary Outcome: Volume of Distribution (Vz/F) of Radiolabelled SSP-004184
Description: The distribution of a medication between plasma and the rest of the body.
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
Liters | 216.534 (57.590)

7. Primary Outcome: AUC 0→∞ Whole Blood Total Radioactivity of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: ng equivalents*hr/g
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
ng equivalents*hr/g | 156702.7 (18867.3)

8. Primary Outcome: Cmax Whole Blood Total Radioactivity of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: ng equivalents/ml
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
ng equivalents/ml | 57216.7 (15434.7)

9. Primary Outcome: Tmax Whole Blood Total Radioactivity of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Median (Full Range); unit: hours
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
hours | 1.5 [1.0 to 1.5]

10. Primary Outcome: Half-Life Whole Blood Total Radioactivity of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
hours | 2.863 (1.687)

11. Primary Outcome: CL/F Whole Blood Total Radioactivity of Radio-Labelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
L/hr | 19.396 (2.623)

12. Primary Outcome: Vz/F Whole Blood Total Radioactivity of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
Liters | 76.731 (39.114)

13. Primary Outcome: AUC 0→∞ Plasma Total Radioactivity of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: ng equivalents*hr/ml
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
ng equivalents*hr/ml | 293626.3 (78627.1)

14. Primary Outcome: Cmax Plasma Total Radioactivity of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: ng equivalents/ml
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
ng equivalents/ml | 103650.0 (29083.6)

15. Primary Outcome: Tmax Plasma Total Radioactivity of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Median (Full Range); unit: hours
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
hours | 1.5 [1.0 to 1.5]

16. Primary Outcome: Half-Life Plasma Total Radioactivity of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
hours | 9.389 (3.538)

17. Primary Outcome: CL/F Plasma Total Radioactivity of Radio-Labelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
L/hr | 11.071 (3.947)

18. Primary Outcome: Vz/F Plasma Total Radioactivity of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
Liters | 137.108 (23.637)

19. Primary Outcome: Percent Total Radioactivity Excreted in Urine of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: percentage of radioactivity
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
percentage of radioactivity | 62.4 (14.5)

20. Primary Outcome: Percent Total Radioactivity Excreted in Stool of Radiolabelled SSP-004184
Time Frame: as for outcome 1
Population: PAS
Measure: Mean (Standard Deviation); unit: percentage of radioactivity
Arm/Group | [14C]SSP-004184
Number analyzed (Participants) | 6
percentage of radioactivity | 29.9 (13.2)

ADVERSE EVENTS:
Arm/Group | [14C]SSP-004184
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [14C]SSP-004184 (N=6)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Chromaturia (Renal and urinary disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.